CLINICAL TRIAL: NCT04767204
Title: The Factors Related to Occupational Outcome Among Persons With Mental Illness Under the Peer-support Service in Vocational Rehabilitation Program: a Pilot Study
Brief Title: The Outcomes Among Persons With Schizophrenia Under the Peer-support Service in Vocational Rehabilitation Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yu-Li Hospital (Other)
Collaborators: Workforce Development Agency of Minister of Labor, Taiwan (Unknown); Tzu-Chi University, Department of Public Health (Unknown); Taipei Veterans General Hospital Yuli Branch, Department of Psychiatry (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: VHYL-107-11
Record Dates: First submitted 2021-02-08; First posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Schizophrenia
Keywords: Peer support; Vocational rehabilitation; Social function
MeSH Terms: conditions — Schizophrenia; Social Adjustment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peer support service (Experimental): Peer support workers co-lead and assist workplace problem-solving and care skills training in an extended vocational rehabilitation program
  Interventions: Behavioral: peer co-delivered vocational rehabilitation service

INTERVENTIONS:
Behavioral: peer co-delivered vocational rehabilitation service — The services provided by the trained peers in the work training or problem-solving group, which integrates into a supported employment services
  Other Names: vocational peer support service

SUMMARY:
There are few programs related to vocational peer support services in persons with psychiatric disability in Taiwan. This study aims to develop a peer co-lead services in the community rehabilitation center and evaluate the outcomes among service users with schizophrenia under the integrated peer-support services in a supported employment program.

DETAILED DESCRIPTION:
Background

In Taiwan, mental health services are provisioned through hospital-based treatment majorly and shifted to community care gradually in recent decades. In 2020, the totally 7,350 beds of acute wards and 13,559 beds of chronic wards covered the general population in Taiwan with 3.12/10,000 persons and 5.75/10,000 persons rates, respectively. In contrast to hospital treatment, there were 71 community rehabilitation centers and 155 halfway houses in local communities with coverage rate of 1.45/10,000 persons and 2.82/10,000 persons respectively. The sheltered or supported employment in Taiwan is still primarily delivered by trained professionals or paraprofessionals in the community facilities for the persons with severe mental illness. Although the trained peers can deliver vocational supports based on recovery concept as well as professionals at least in the supported employment services, the large absence of peer support workers is rooted in the lack of insurance coverage and limited government budgets in Taiwan. Accordingly, further investigations are warranted to evaluate the effectiveness of peer support services in vocational rehabilitation among persons with severe mental illness under the development of peer-deliver services in Taiwan.

Therefore, the investigators designed a 2-phase pilot program: establishment of peer support training curriculum in Phase I to develop peer support services in vocational rehabilitation system feasibly, and measurement of effectiveness under peer codelivered services in Phase II (Protocol). The investigated effectiveness among persons with schizophrenia in this study included the received social supports, mental health, psychiatric symptoms, functional and occupational outcome.

Methods

Participants

The pilot program was held from April 2017 to December 2018 at the Taipei Veterans General Hospital Yuli Branch (TVGH-YL). The hospital provides treatment and community care for patients with mental illness who reside in the rural area of eastern Taiwan. The TVGH-YL administers a half-way house, a community rehabilitation center, and a supported housing program. The hospital also provides sheltered and supported employment as part of its community care services for persons with mental illness. In one month before the program of Phase I or II, the investigators recruited the participants by presenting poster on bulletins in the half-way house and community rehabilitation center. The investigators also invited the participants who had cared elderly persons in the past to join the training curriculum in the Phase I program, because these persons were the candidates of peer support workers to share the previous work experiences in the Phase II program.

Pilot program

Training for peer support workers

Initially, there were 7 professionals who had the experiences in the community facilities for at least 5 years discussing about the framework and contents of training curriculum for peer support workers in the focus groups. These seven professionals specializing in 6 medical disciplines were also the teachers in the curriculum. Table 2 details the themes of curriculum at various intervention levels. In the end of each lecture session, there were four questions being proposed by the teacher to exam the trainees about the core concepts of class.

In the practice session, the performance of trainees would be examined by the case discussion or practice in roles playing or situation simulation. No final exam in Phase I program. However, the trainee should pass all class after the teachers' agreement. If someone needed to improve the knowledge or skills, he or she had gotten the personal time to receive more helps from the teacher.

The extended vocational rehabilitation services co-led & assisted by peer support workers

The program in Phase II was held twice in August of 2017 and April of 2018. Based on the needs of elderly persons with disability or dementia in local community, the 2 occupational therapists (Ching-Hui Wu & Meng-Ping Kao) organized the extended work training course which focused on improvements of care skills of Phase II program participants (service users). The 2 occupational therapists also held workplace problem-solving group once per 2 weeks for the service users. The above interventions were originally parts of supported employment service in the community rehabilitation center, but the participated rate was not satisfied previously. Therefore, the investigators integrated the peer support service into this service system. Before each training session, peer support workers discussed with 2 occupational therapists ("stakeholders") to decide on the content and process of the session. Peer support workers' involvement should account for at least 50% of the session time to ensure the intensity of support. The supervisor (Kan Yuan Cheng) discussed with the occupational therapy weekly and the peer support worker monthly based on the feedback in satisfaction questionnaire by service users and the records in group. Four times of observation by the supervision were also arranged to audit the performance of the occupational therapist and peer support workers in the all sessions of Phase II program. More specifics about this phase of the program can be found in study protocol.

Process of assessment

The pre- and post-intervention self-report questionnaire was assisted by the occupational therapist ( Meng-Ping Kao). The Brief Psychiatric Rating Scale-18 and Global Assessment of Function scale were measured by board psychiatrist (Kan Yuan Cheng) who had experiences in the multiple-center clinical trial. The assistant and investigator both belonged to the intervention group because there was no control group or blind procedure in the study design.

Statistical methods

As all indicators examined in this study were continuous variables, the investigators used paired t-test to compare the measurements before and after the intervention. IBM (International Business Machines Corporation) SPSS Statistics 16.0 was employed for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnoses of schizophrenia
* Living in half-way houses or community home
* Under the services of sheltered or supported employment
* The reading ability of graduated elementary school at least

Exclusion Criteria:

* Acute psychosis
* Severe physical illness
* Legally incompetence to make major decision

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-09-28 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Change of Social Support Scale | Changes from Baseline Social Support Scale at 4 months
  SSS. Social supports from family or relatives, professionals or staffs and peers or friends. Ranges from 45 to 225. Higher score means better support.
Change of Chinese Health Questionnaire-12 | Change from Baseline Chinese Health Questionnaire-12 at 4 months
  CHQ-12. Positive and Negative Mental health. Ranges from 0 to 12. Lower score means better health.
Change of Brief Psychiatric Rating Scale-18 | Change from Baseline Brief Psychiatric Rating Scale-18 at 4 months
  BPRS-18. Mood, Psychotic and General symptoms. Ranges from 18 to 126. Higher score means worse psychiatric symptom.
Change of Global Assessment of Function | Change from Baseline Global Assessment of Function at 4 months
  GAF. Globally social and occupational function under the influences by the mental illness. Ranges from 1 to 100. Higher score means better function.
Change of Chinese version of the Social Functioning Scale | Change from Baseline Chinese version of the Social Functioning Scale at 4 months
  C-SFS. Self-reported social function for the persons with schizophrenia. Ranges from 0 to 100. Higher score means better function

SECONDARY OUTCOMES:
Change of weekly wedges | Change from Baseline weekly wedges at 4 months
  totally earned incomes through the vocational rehabilitation services
Change of weekly working hours | Change from Baseline weekly working hours at 4 months
  totally working hours through the vocational rehabilitation services

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital Yuli Branch, Yuli, Haulein County, Taiwan

IPD SHARING:
Plan to Share IPD: No
Any share of data related to persons with mental illness in Taiwan should be permitted by the Institute Review Board. Under the asking of IRB, we must destroyed any kinds of study data when three years after completed collection. This requirement was also described in the informed consent.

REFERENCES:
- [Background] Lloyd-Evans B, Mayo-Wilson E, Harrison B, Istead H, Brown E, Pilling S, Johnson S, Kendall T. A systematic review and meta-analysis of randomised controlled trials of peer support for people with severe mental illness. BMC Psychiatry. 2014 Feb 14;14:39. doi: 10.1186/1471-244X-14-39. PMID 24528545
- [Background] Yam KKN, Lo WTL, Chiu RLP, Lau BSY, Lau CKS, Wu JKY, Wan SM. A pilot training program for people in recovery of mental illness as vocational peer support workers in Hong Kong - Job Buddies Training Program (JBTP): A preliminary finding. Asian J Psychiatr. 2018 Jun;35:132-140. doi: 10.1016/j.ajp.2016.10.002. Epub 2016 Oct 24. PMID 27884479
- [Background] Kern RS, Zarate R, Glynn SM, Turner LR, Smith KM, Mitchell SS, Becker DR, Drake RE, Kopelowicz A, Tovey W, Liberman RP. A demonstration project involving peers as providers of evidence-based, supported employment services. Psychiatr Rehabil J. 2013 Jun;36(2):99-107. doi: 10.1037/h0094987. PMID 23750760
- [Derived] Cheng KY, Yen CF. The social support, mental health, psychiatric symptoms, and functioning of persons with schizophrenia participating in peer co-delivered vocational rehabilitation: a pilot study in Taiwan. BMC Psychiatry. 2021 May 25;21(1):268. doi: 10.1186/s12888-021-03277-0. PMID 34034693